CLINICAL TRIAL: NCT01676987
Title: Evaluation of the Efficacy and Safety of a Fixed-dose, Single-capsule Budesonide-formoterol Combination in Uncontrolled Asthma:a Randomized, Double-blind, Multicenter, Controlled Clinical Trial.
Brief Title: Evaluation of the Efficacy and Safety of a Fixed-dose, Single-capsule Budesonide-formoterol Combination in Uncontrolled Asthma
Acronym: Ach-ALN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ach-ALN-04(7/07)
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Asthma
Keywords: Asthma; Budesonide; Adrenergic beta-2 receptor agonists.
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fixed Combination of Budesonide and formoterol (Experimental): Group 1 (experimental): Fixed Combination of Budesonide and formoterol
  Interventions: Drug: Fixed combination of budesonide and formoterol
- Budesonide (Active Comparator): Group 2 (comparator): Budesonide
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Fixed combination of budesonide and formoterol — Delivered dry powder inhaler for 12 weeks.
  Other Names: Group 1 (experimental): Budesonide and formoterol
  Arms: Fixed Combination of Budesonide and formoterol
Drug: Budesonide — Delivered dry powder inhaler for 12 weeks.
  Other Names: Group 2 (comparator): Budesonide
  Arms: Budesonide

SUMMARY:
To evaluate the efficacy and safety of a fixed-dose, single-capsule budesonide(400µg)-formoterol(12µg) combination, in comparison with budesonide alone, both delivered via a dry powder inhaler, in 181 patients with uncontrolled asthma.This was Randomized, double-blind, multicenter, phase III, parallel clinical trial.

DETAILED DESCRIPTION:
the age of the patients ranged from 18 to 77 years. After a run-in period of 4 weeks, during which all of the patients received budesonide twice a day, they were randomized into one of the treatment groups for 12 weeks, twice a day.

The primary outcome measures were FEV1, FVC and morning PEF. We performed an intention-to-treat analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of uncontrolled asthma
* Age ranged from 18 to 77 years
* Nonsmokers

Exclusion Criteria:

* Use of oral corticosteroids, anti-leukotrienes, immunoglobulins, beta blockers, digitalis, amiodarone, antifungals, antidepressants, monoamine oxidase inhibitors and tricyclics during the standardization
* Atrial fibrillation, Flutter, severe and complex tachyarrhythmias atrioventricular block 1,2 and 3
* Diabetes mellitus
* Pregnancy
* Neuropsychiatric diseases
* Pulmonary malformations, tuberculosis, Cystic fibrosis
* Immunosuppressive treatment
* Hospitalization for asthma or respiratory infection in last 30 days
* Severe systemic disease

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy and safety of a fixed-dose, single capsule budesonide-formoterol combination in comparison with budesonide alone in patients with uncontrolled asthma | 12 weeks
  the primary outcome Measures were FEV1(forced expiratory volume in one second), FVC(forced vital capacity)and morning PEF (peak expiratory flow).

CONTACTS AND LOCATIONS:
Overall Officials: Emílio Pizzichini, Principal Investigator — NUPAIVA Asthma Research Center, UFSC- Brazil

REFERENCES:
- [Derived] Stirbulov R, Fritscher CC, Pizzichini E, Pizzichini MM. Evaluation of the efficacy and safety of a fixed-dose, single-capsule budesonide-formoterol combination in uncontrolled asthma: a randomized, double-blind, multicenter, controlled clinical trial. J Bras Pneumol. 2012 Jul-Aug;38(4):431-7. doi: 10.1590/s1806-37132012000400004. English, Portuguese. PMID 22964926